CLINICAL TRIAL: NCT06020833
Title: A Single-arm Trial of Roxadustat Combined With Retinoic Acid in the Treatment of Refractory Low-risk MDS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Roxadustat-RA-MDS
Record Dates: First submitted 2022-02-17; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — roxadustat; Tretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Roxadustat combined with retinoic acid group (Experimental)
  Interventions: Drug: Roxadustat in combination with retinoic acid

INTERVENTIONS:
Drug: Roxadustat in combination with retinoic acid — Roxadustat 150mg po qod combined with retinoic acid 20mg po bid

SUMMARY:
Roxadustat has been approved for low-risk MDS clinical trials, but the trial results are not available. For refractory low-risk MDS, the effective rate of roxadustat treatment is about 20-30%, and roxadustat combined with retinoic acid may have better efficacy in the treatment of refractory low-risk MDS.

DETAILED DESCRIPTION:
Patients with low-risk myelodysplastic syndrome who are refractory to the regular treatments have to live on transfusions which lead to poor quality of life (QoL) and survival. Roxadustat, an oral hypoxia-inducible factor prolyl hydroxylase inhibitor, which increases both endogenous EPO and iron metabolism, has shown promising results in several phase 3 clinical trials for chronic kidney disease.

Roxadustat comprehensively improves iron metabolism by upregulating DCYTB and DMT1 through the HIF pathway, which can promote the iron absorption and utilization. Detail mechanisms include upregulating transferrin receptors to increase iron uptake, upregulating transferrin to promote iron transport and downregulating ferritin levels to indirectly improve iron absorption and transportation.

Patients with refractory low-risk MDS were selected and given roxadustat 150mg po qod combined with retinoic acid 20mg po bid.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk MDS unresponsive to first-line therapy

Exclusion Criteria:

* myelofibrosis
* Severe heart and kidney function bu'quan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (OR) | 3, 6 months
  Complete and partial remission with roxadustat combined with retinoic acid. Partial remission includes freedom from transfusion dependence or reduction in transfusion volume within 8 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carraway HE, Saygin C. Therapy for lower-risk MDS. Hematology Am Soc Hematol Educ Program. 2020 Dec 4;2020(1):426-433. doi: 10.1182/hematology.2020000127. PMID 33275714